CLINICAL TRIAL: NCT06499077
Title: Non-invasive Detection of Breast Cancer by Mass-spectrometry-based Profiling of Exhaled Breath
Brief Title: Non-invasive Detection of Breast Cancer by Breath Analysis
Acronym: BreathBC
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: IstitutoTumori-BreathBC
Record Dates: First submitted 2024-06-04; First posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-05

CONDITIONS: Breast Neoplasm Female
Keywords: breath analysis; non invasive detection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tumor: Women carrying a breast cancer
  Interventions: Diagnostic Test: Sampling of exhaled breath
- Control: Women with negative breast imaging
  Interventions: Diagnostic Test: Sampling of exhaled breath

INTERVENTIONS:
Diagnostic Test: Sampling of exhaled breath — Exhaled breath of all participants is collected following our standardized procedure

SUMMARY:
The goal of this prospective observational study is to compare the exhaled breath profiles of patient with invasive breast cancer and control subjects in the perspective of a diagnostic application in oncology.

The main question it aims to answer is whether the exhaled breath profile of breast cancer patients can be discriminate from the exhaled breath of control subjects.

Participants to the study are recruited in a first discovery series including about 500 subjects and in a following independent validation series including more than 400 subjects. Breath samples are collected in a dedicated room using sampling bags and following anti-Covid-19 measures. Only authorized personnel could access the sampling room which was equipped with a HEPA Filter air purification system. Sampling bags are made of Nalophan® tubular foil and 2 taps, one in which the study participant inflated with their breath and sealed after use, while the second is used to introduce breath samples into the analyzer. Bags are sterilized with the Sterrad™ system with H2O2 vapors before use. To contain the potentially infectious particulate included in the participant exhaled breath, an electrostatic filter is mounted on the tap of the bag used to inflate it with breath. All participants are supplied with a leaflet explaining aims and technical/clinical information of the study. At each breath sampling, study participants are asked not to smoke, eat, drink (except for water), brush their teeth or use lipstick for at least 2 h before breath collection to minimize the presence of contaminant molecules in exhaled breath.

Breath profiling is performed by mass spectrometry analysis using an untargeted approach. Breath samples are profiled by Secondary Electrospray ionization - High resolution Mass Spectrometry (SESI-HR-MS) using a high resolution instrumentation (LTQ Orbitrap Elite,Thermo Fisher Scientific) equipped with a SuperSESI ionization source (Fossiliontech).

Data analysis is based on our previous work (Martínez-Lozano el al., 2015 J Breath Res 9:031001) and will be implemented with machine learning and other Artificial Intelligence (AI) methods.

Once all the breath profiles will be collected and analysed, researchers will compare data from patient with breast cancer and data from tumor-free subjects to identify methods and patterns able to specifically identify the pathological breath samples and discriminate them from the control breath samples.

ELIGIBILITY:
Inclusion Criteria:

1. be >= 18 years
2. Patients

2.a patients at early stage of breast cancer 2.b exahled breath collected and analysed at the baseline before any surgical or pharmacological treatment

3. Controls 3.1 subjects with negative breast imaging (BI-RADS= 1,2) 3.2 exhaled breath collected and analysed on the day of breast screening

-

Exclusion Criteria:

1. any cancer in the 5 years before the inclusion
2. major surgery within 4 weeks before the inclusion
3. previous or concomitant long-term treatment with systemic steroids or immunosuppressive/immunomodulating drugs
4. concomitant acute infection, viral hepatitis, HIV infection, COVID19 infection or other serious concomitant medical disorders
5. organ allograft

   -

Ages: 18 Years to 98 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are recruited at Breast Surgery unit of Fondazione IRCCS Istituto Nazionale Tumori in Milan.
  Controls are recruited during breast screening at Breast Imaging Unit of Fondazione IRCCS Istituto Nazionale Tumori in Milan.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Classification of the exhaled breath of breast cancer patients and controls as assessed by the comparison of the global breath profile of volatile organic compounds (VOCs) measured using Mass Spectrometry analysis. | Breath collection and MS analysis were assessed at the baseline.
  Breath profile of each study participant was determined by Mass Spectrometry analysis (Secondary Electrospray ionization - High resolution Mass Spectrometry, SESI-HR-MS). The risk of cancer is identified in the validation cohort of the present study and is based on the diagnostic model developed in the discovery phase of the same study. The predictive result is compared, in the case of breast cancer patients, with the histopathological proven diagnosis and, in the case of control subjects, with the imaging proven diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Rosaria Orlandi, Principal Investigator — Fondazione IRCCS ISTITUTO NAZIONALE TUMORI
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martinez-Lozano Sinues P, Landoni E, Miceli R, Dibari VF, Dugo M, Agresti R, Tagliabue E, Cristoni S, Orlandi R. Secondary electrospray ionization-mass spectrometry and a novel statistical bioinformatic approach identifies a cancer-related profile in exhaled breath of breast cancer patients: a pilot study. J Breath Res. 2015 Sep 21;9(3):031001. doi: 10.1088/1752-7155/9/3/031001. PMID 26390050